CLINICAL TRIAL: NCT05561842
Title: Tablet-based Mobile Health Ultrasound for Point-of-care Breast Cancer Diagnosis in Nigeria
Brief Title: Tablet-based Mobile Health Ultrasound for Point-of-care Breast Cancer Diagnosis in Nigeria (Mobile Health: Technology and Outcomes in Low and Middle-Income Countries)
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-325
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: breast ultrasound; breast cancer; breast biopsy; breast cancer diagnosis; 21-325; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with a solid mass on breast ultrasound: Participants will have a solid mass on breast ultrasound that is suspicious for breast cancer.
  Interventions: Procedure: mHealth US-breast biopsy

INTERVENTIONS:
Procedure: mHealth US-breast biopsy — During this study, women will undergo an US-guided breast biopsy by a radiologist instead of what is typically performed in Nigerian hospitals, which is either a blind biopsy or surgical excision. US-guided breast biopsy is the standard of care in the United States of America because the accuracy is better than blind biopsy and equal to surgical excision.

SUMMARY:
The purpose of this study is to train Nigerian radiologists to perform ultrasound-guided breast biopsies. Researchers will use mHealth devices to create a sustainable and practical way of training radiologists in Nigeria to perform and clinically implement US-guided breast biopsies into their practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older female.
* Breast ultrasound demonstrating a solid mass that is suspicious for cancer, which would typically undergo either a blind biopsy or surgical excision at the Nigerian hospital where the patient is seeking diagnosis.

Exclusion Criteria:

* Participants unwilling to sign consent.
* Participants under the age of 18.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be accrued in medical clinics as determined by the local investigators and local research staff. Informed consent forms approved by each local IRB will be obtained by research staff from each site.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2027-09-21 (Estimated)

PRIMARY OUTCOMES:
Number of successful US-guided breast biopsy | 1 year
  Trainees will be evaluated using a passing criterion of 80% on a validated test that assesses competency based on the The Ottawa Surgical Competency Operating Room Evaluation (O-Score). There are 8 variables rated on a scale of 1-5. A trainee will be given a passing grade if the responses on all 8 variables are 4 or 5 and this is achieved in at least 80% of the unsupervised simulation and patient biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Eliabeth Sutton, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States
- Nigeria (7):
  - Lagos University Teaching Hospital, Idi Araba, Lagos
  - Olabisis Onabanjo University Teaching Hospital (Data Collection Only), Sagamu, Ogun State
  - Federal Medical Centre Owo (Data Collection Only), Owo, Ondo State
  - University College Hospital (Data Collection Only), Ibadan, Oyo State
  - University Of Nigeria Teaching Hospital (UNTH) Ituku-Ozalla Enugu, Enugu
  - Obafemi Awolowo University Teaching Hospitals Complex (Data Collection Only), Ile-Ife
  - University of Ilorin Teaching Hospitals, Ilorin

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org